CLINICAL TRIAL: NCT03029715
Title: Comparative Study Between Inhalational Anaesthesia and Total Intravenous Anaesthesia (TIVA) With Dexmedetomidine for Morbidly Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Anaesthesia for Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dr Ezzeldin Ibrahim, Assistant Professor in anaesthesia, intensive care, and pain medicine., Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MenoufiaU2016/2
Record Dates: First submitted 2017-01-14; First posted 2017-01-24 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Obese
Keywords: Sleeve gastrectomy; TIVA
MeSH Terms: conditions — Obesity | interventions — Propofol; Remifentanil; Dexmedetomidine; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous anaesthesia (Other): Propofol Dexmedetomidine Remifentanil
  Interventions: Drug: Propofol; Drug: Remifentanil; Drug: Dexmedetomidine
- Inhalation anaesthesia (Other): Desflurane Remifentanil
  Interventions: Drug: Remifentanil; Drug: Desflurane

INTERVENTIONS:
Drug: Propofol — Total intravenous anaesthesia.
  Other Names: TIVA group
  Arms: Intravenous anaesthesia
Drug: Remifentanil — Narcotics
  Other Names: TIVA group and inhalation group
Drug: Dexmedetomidine — Total intravenous anaesthesia
  Other Names: TIVA group
  Arms: Intravenous anaesthesia
Drug: Desflurane — Inhalation anaesthesia.
  Other Names: Inhalation group
  Arms: Inhalation anaesthesia

SUMMARY:
Background: Laparoscopic sleeve gastrectomy is commonly done with total intravenous anaesthesia (TIVA) or balanced anaesthesia using intravenous and an inhalation agent. It is still unclear which anaesthesia regimen is better for this group of patients. The present study was carried out to compare the use of inhalation anaesthesia technique using desflurane and TIVA using propofol and dexmedetomidine.

Methods: This randomized controlled trial was carried out on 100 morbidly obese patients undergoing laparoscopic sleeve gastrectomy. The patients were randomized into two equal groups, inhalational group and TIVA group for anaesthesia maintenance. All patients received general anaesthesia and induced with propofol, remifentanil and cis-atracurium. In inhalation group, anaesthesia was maintained by desflurane in oxygen air mixture while in TIVA group anaesthesia was maintained by intravenous propofol and dexmedetomidine infusion. Intra-operative vital signs and anaesthesia recovery time were recorded. Post-operative nausea, vomiting, pain score, analgesic consumption, the onset of bowel movement, and post-anaesthetic care unit (PACU) stay were studied for both groups.

DETAILED DESCRIPTION:
After obtaining the ethics committee approval of El Menoufia University hospital and the informed written consent from the patients, a hundred morbidly obese patients scheduled for sleeve gastrectomy were recruited for the study. Patients with history of cardiac comorbidity, chronic obstructive lung disease, drug abuse, expected difficult intubation patients, and patients with history of allergy to the study drugs were excluded from the study. Patients from 30 to 50 years old of both sexes were randomly allocated using computerized software into two groups, fifty patients in each group. Patients in inhalation group received intra-operative inhalational anaesthetic while patients in TIVA group received TIVA for anaesthetic maintenance.

All patients received a routine premedication with oral sodium citrate 15ml [0.3 molar (1.16gm)] and intravenous (IV) 4mg ondansetron fifteen minutes before induction. Patients in both groups were connected to the routine monitoring and bispectral index (BIS) upon arrival to theatre. Anaesthesia induction for both groups was carried out by 0.5-1 mcg kg -1 remifentanil, 2-3mg kg-1 propofol, and 0.6 mg kg-1 rocuronium. Endotracheal intubation was done with the appropriate tube size.

In the inhalational group, anaesthesia was maintained by desflurane in low flow oxygen air mixture 60/40%. In the TIVA group, anaesthesia was maintained using propofol 8-12 mg kg-1 h-1 and dexmedetomidine 0.5-1ugkg-1h-1. Remifentanil infusion of 0.05-2 µg kg-¹min-¹ was administered for both groups. Muscle relaxation was maintained in both groups by rocuronium infusion at a rate of 10-12ug kg1min-1. Depth of anaesthesia was monitored by bispectral index and anaesthetics were adjusted in both groups to obtain BIS of 40 to 60 by giving boluses of 0.5ug kg-1 remifentanil. The total boluses of intra-operative remifentanil were recorded. At the end of the procedure all patients received 0.6mg atropine and sugammadex 16mg kg-1 to reverse the effect of rocuronium. Patients were extubated and transferred to the post-anaesthetic care unit (PACU).

Post-operative pain was monitored using visual analogue score (VAS) at PACU. Morphine sulphate 2 to 3 mg was given if the VAS was > 4. Intravenous paracetamol 1gm and/or ketorolac 30 mg were given eight hourly intravenously if needed (VAS ≥3). Post-operative ondansetron 4mg every eight hours was given if required.

Haemodynamics including heart rate and mean arterial blood pressure (MABP) were recorded as a baseline and every fifteen minutes intra-operatively. Recovery time from anaesthesia using Aldrete score was recorded (the time from cessation of all anesthetics until complete recovery). 10 The incidence of post-operative nausea and vomiting, post-operative analgesic requirements, and the duration of PACU stay were recorded. Post-operative pain assessment using VAS from 0 to 10, where 0 means no pain and 10 is the worst pain the patient experienced. VAS was recorded at full recovery, every 15 minutes in PACU until discharge PACU. Time of onset of post-operative bowel movement was recorded.

Statistical analysis:

Sample size calculation was calculated using Graphed Instant statistics version 3. Based on the previous, studies propofol was expected to produce a drop in the MABP after induction of anaesthesia by about 10 mmHg with a standard deviation of 15 mmHg so by choosing level of significance 0.05 and power of 90%; the calculated sample size was 48 patients so that the number of patients randomized in each group was fifty patients to ensure reliable results.

Statistical analysis was done using SPSS 19 (SPSS Inc, IBM company, Chicago,USA). The patients' sex, American society of anaesthetists (ASA) status and incidence of side effects were analyzed using the chi-square χ2-test. Other parameters were compared using student t-test. For comparisons within the same group, paired t-test was used where for comparisons between groups; unpaired t-test was used. P-value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese scheduled for sleeve gastrectomy.

Exclusion Criteria:

* Patients refusal and allergy to drugs used.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elbakry AE, Sultan WE, Ibrahim E. A comparison between inhalational (Desflurane) and total intravenous anaesthesia (Propofol and dexmedetomidine) in improving postoperative recovery for morbidly obese patients undergoing laparoscopic sleeve gastrectomy: A double-blinded randomised controlled trial. J Clin Anesth. 2018 Mar;45:6-11. doi: 10.1016/j.jclinane.2017.12.001. Epub 2017 Dec 8. PMID 29223575

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Anaesthesia | Inhalation Anaesthesia
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Anaesthesia | Inhalation Anaesthesia | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.31 (10.43) | 34.35 (11.15) | 34.83 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 33 | 68
  Male | 15 | 17 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Analgesic Requirements.
Description: Total paracetamol consumption.
Time Frame: Within one hour after surgery
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Sleeve Gastrectomy 1: Propofol Dexmedetomidine Remifentanil
  Propofol: Total intravenous anaesthesia.
  Remifentanil: Narcotics
  Dexmedetomidine: Total intravenous anaesthesia
- Sleeve Gastrectomy 2: Desflurane Remifentanil
  Remifentanil: Narcotics
  Desflurane: Inhalation anaesthesia.
Arm/Group | Sleeve Gastrectomy 1 | Sleeve Gastrectomy 2
Number analyzed (Participants) | 50 | 50
mg | 3.56 (1.01) | 1.67 (1.03)

2. Secondary Outcome: The Intra-operative Mean Arterial Blood Pressure.
Time Frame: During operation and follow-up, an average of 2 hours
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sleeve Gastrectomy 1 | Sleeve Gastrectomy 2
Number analyzed (Participants) | 50 | 50
mmHg | 71.05 (3.06) | 62.7 (2.98)

ADVERSE EVENTS:
Time Frame: During operation and follow-up, an average of 2 hours
Description: Nausea and vomiting
Arm/Group | Intravenous Anaesthesia | Inhalation Anaesthesia
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes